CLINICAL TRIAL: NCT06144372
Title: Comparison of Efficacy and Safety of Extracorporeal Shockwave Lithotripsy: A Randomized, Controlled Trial Study of Electroconductive and Electrohydraulic Types
Brief Title: Extracorporeal Shockwave Lithotripsy, Electroconductive and Electrohydraulic Types
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Cho, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESWL_ECEH
Record Dates: First submitted 2023-11-09; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Urolithiasis
Keywords: Extracorporeal shockwave lithotripsy; Urolithiasis; Radiation Exposure
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroconductive Type (Other): Sonolith i-move® shockwave lithotripter (EDAP, Lyon, France)
  Interventions: Device: Electroconductive and Electrohydraulic types
- Electrohydraulic Type (Other): Rifle lithotripter (HNT Medical, Seoul, Korea)
  Interventions: Device: Electroconductive and Electrohydraulic types

INTERVENTIONS:
Device: Electroconductive and Electrohydraulic types — The patients were randomly assigned to two types of lithotripter.

SUMMARY:
To evaluate the efficacy and safety of electroconductive (EC) and electrohydraulic (EH) extracorporeal shock wave lithotripsy (ESWL) for the treatment of ureter and kidney stones, this study conducted a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* The analysis included cases of stones in the upper kidney and ureter, with diameters ranging from 5 mm to 15 mm.

Exclusion Criteria:

* Patients with musculoskeletal deformities, ongoing urinary tract infections requiring prioritized infection treatment, blood clotting disorders, and ureteral obstruction that made stone expulsion difficult were excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
age | 2 weeks
  patient's records
Gender | 2 weeks
  patient's records
height | 2 weeks
  meters
weight | 2 weeks
  kilograms
smoking | 2 weeks
  patient's records
drinking | 2 weeks
  patient's records
Diabetes mellitus | 2 weeks
  patient's records
Hypertension | 2 weeks
  patient's records
Preoperative Double J stent | 2 weeks
  patient's records
creatinine | 2 weeks
  patient's records
Glomerular Filtration Rate | 2 weeks
  patient's records
hemoglobin | 2 weeks
  patient's records
Hydronephrosis grade | 2 weeks
  * Grade 0 : Normal examination with no dilation of the renal pelvis
  * Grade 1 : Mild dilation of the renal pelvis only
  * Grade II : Moderate dilation of the renal pelvis including a few calyces
  * Grade III : Dilation of the renal pelvis with visualization of all the calyces, which are uniformly dilated, and normal renal parenchyma
  * Grade IV : Similar apperance of the renal pelvis and calyces as Grade III, plus thinning of the renal parenchyma
Analgesic | 2 weeks
  patient's records
stone size | 2 weeks
  patient's records
Stone laterality | 2 weeks
  patient's records
Stone location | 2 weeks
  patient's records
Stone volume | 2 weeks
  patient's records
Stone shape | 2 weeks
  patient's records
Stone to skin distance | 2 weeks
  patient's records
Hounsfield unit | 2 weeks
  patient's records
Urine color | 2 weeks
  patient's records
Urine Turbidity | 2 weeks
  patient's records
Urine Specific Gravity | 2 weeks
  patient's records
Urine pH | 2 weeks
  patient's records
Intensity | 2 weeks
  ESWL
Used power | 2 weeks
  ESWL
Shock | 2 weeks
  ESWL
Speed | 2 weeks
  ESWL
Visual analog scale for pain | 2 weeks
  0: Represents "No sensation" or "Not at all." 1-3: Indicates a very mild sensation or a low level of the experience, signifying almost no problem.
  4-6: Represents a moderate level, suggesting a moderate presence of the experience or issue.
  7-9: Reflects a high or severe level, signifying a significant presence or seriousness of the problem.
  10: Represents "Maximal sensation" or "Extremely intense" and indicates an extreme presence or severity of the experience or issue.
Satisfaction score | 2 weeks
  1. Not satisfied at all.
  2. Very low satisfaction.
  3. Moderate satisfaction.
  4. High satisfaction.
  5. Very high or maximum satisfaction.
Stone-free rates (%) | 2 weeks
  ESWL

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The datasets used during the current study are available from the corresponding author on request.

REFERENCES:
- [Background] Motolova M, Kral M. Effect of targeting and generator type on efficacy of extracorporeal shock wave lithotripsy. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2022 Dec;166(4):434-440. doi: 10.5507/bp.2022.029. Epub 2022 Jun 27. PMID 35801399